CLINICAL TRIAL: NCT02480179
Title: CNS Modification of Food Craving by Neurofeedback
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Ruth Perchik, Dr., Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1164-14-SMC
Record Dates: First submitted 2015-05-28; First posted 2015-06-24 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Obesity
Keywords: functional MRI; appetite; neurofeedback
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single arm pilot feasibility study (Experimental): Hematoencephalography bio/neurofeedback for Brain neural activity modulation. H.E.G. (hematoencephalography) based neurofeedback program. No drug use.
  Interventions: Device: H.E.G. (hematoencephalography) based neurofeedback

INTERVENTIONS:
Device: H.E.G. (hematoencephalography) based neurofeedback — H.E.G. is a relatively new neurofeedback technique which, similar to fMRI is based on differential oxygenated blood supply according to regional brain activity.
  Other Names: ProComp2 - 2 Channel Biofeedback & Neurofeedback System w/ BioGraph Infiniti Software - T7400M

SUMMARY:
The investigators plan to evaluate H.E.G. (Hematoencephalography) modality in brain modulation of appetite and food craving in a randomized controlled study. The H.E.G. will serve as the neurofeedback modality while the functional brain imaging will enable assessment and hopefully validation of changes brain activity related to food craving and self-control. H.E.G. is a relatively new neurofeedback technique which similar to fMRI, is based on changes in blood oxygenation level as a result of regional brain activation. The unique advantage of this technology regarding our enterprise is that it inheritably samples the two brain areas that are in our focus of interest: the superior orbito-frontal cortex (OFC) which Involved in self-control and reward processing, and the anterior cingulate cortex (ACC) which processes cognitive and emotional information. The investigators will combine HRV (Heart rate variability) biofeedback, which is a well-established treatment form in the investigators therapeutic sessions and will correlate functional neuroimaging with behavioral, anthropometric and laboratory data.

The intervention name is: Measurements of blood flow changes within the brain and online visual feedback to the participant by a H.E.R. (Hematoencephalography) N.I,R (Near Infra Red sensor) sensor made by MindMedia, The Netherlands and a NEXUX4 Hardware, Bluetooth unit, Bio Trace Plus software made by MindMedia, The Netherlands.

Hypothesis: The neurofeedback practice sessions are expected to facilitate improved control of blood flow to frontal brain areas, as a marker of brain activity in these areas

DETAILED DESCRIPTION:
CNS Modification of Food Craving by Neurofeedback Study Protocol Research Plan and Methodology

The investigators's goal is to modulate food craving and eating behavior among overweight and obese participants using and interventional neurofeedback program. During the study period, each participant will go through 10 neurofeedback sessions, two sessions per week, over a five-week period. In addition, each participant will go through two functional MRI sessions, the first session, before the neurofeedback intervention, to document baseline neurocognitive response to food stimuli using a specified paradigm and the second - after completion of the neurofeedback series, in order to evaluate changes in C.N.S. response to food.

Subjects: 6 overweight and obese participants will be participate in our pilot study and will go through 2 fMRI sessions, 10 H.E.G. sessions and 3 anthropometric and metabolic evaluations during one year intervention and follow-up.

Study Design: In the investigators's single arm pilot study participants will go through a series of neurofeedback sessions with psychological, anthropomorphic, and laboratory evaluation taken before and after intervention.

Baseline questioners: Baseline assessment will include completion of a combined questionnaire that will address a spectrum eating behavior traits, including hunger and craving, addiction, impulsivity, binge eating, addiction, impulsivity, hedonic eating and externally driven eating14-23.

Anthropomorphic measurements: Height, weight, waist circumference and BMI will be measured before intervention. Weight and calculated BMI will be documented twice more: at week 7-8, soon after accomplishing the Neurofeedback sessions series and at week 12.

The investigators intend to call participants 6 and 12 months after study start and ask for their current weight.

Blood samples: Gut peptides and hormones that are known to parallel weight changes will be measured in the first and last visits including: leptin, morning cortisol, TSH, Ft4 and TT3. In addition, before each fMRI session we will evaluate "satiety profile" by documenting levels of Ghrelin, PYY, c-peptide and insulin.

Functional MRI sessions Experimental Paradigm Based on current knowledge regarding brain areas involved in food craving, the investigators defined two ROIs (regions of interest) that correspond with the introspective tasks in the H.E.G. neurofeedback sessions, one area in the superior orbitofrontal cortex (sOFC.) bilaterally and the second: the anterior cingulated cortex (ACC) bilaterally. Each ROI will be mapped in a block design paradigm (7:22 min) in which visual food stimuli will be shown alternately with neutral visual stimuli (neutral objects) and fixation (8 cycles, 54sec each including 3 blocks, 18s each of fixation, neutral objects, and food stimuli).

For the investigator's specific modulation goal, the suitable in-scanner satiety status is "half satiated". On one hand, hunger activates brain circuits involved in homeostatic appetite while, on the other hand complete satiety will shut down any food craving. For that purpose, participants will be asked to time their meals in order to start the session 1-2 hours after a medium-large meal. The investigators will document in detail the last meal (timing, content, estimated caloric value) and explore correlative parameters in the hormonal profile. Participants will be asked to rate their hunger, satiety, fullness and prospective eating in visual analogue scales: graphic questioners that are commonly used and well validated in eating behavior research field.

fMRI data acquisition: Functional scanning will be performed using a 3 Tesla whole body MRI system (GE EXITE HDxt, most updated version 14 M5) equipped with 8-channel head coil. Each scan will be acquired using a standard gradient echo planar imaging (EPI) sequence. After each volume is acquired, it will be automatically transferred in DICOM format from the MRI scanner computer to a separate computer for in-scan processing.

fMRI data processing: Online RT-fMRI processing will be made possible via a fast connection between the MRI scanner and the analysis/display computer. Turbo-Brain Voyager (TBV) 2.0 software (Brain Innovation, Maastricht, the Netherlands) will be used to perform real-time in-scan processing. TBV is capable of incrementally computing statistical maps based on General Linear Model (GLM) and event-related averages.

Off-line fMRI analysis:

Off-line analysis will be conducted to all data collected. Off-line analysis will be performed using Statistical Parametric Mapping software 8 (SPM8. The Welcome Department of Cognitive Neurology, London, UK). While MarsBar toolbox (the Marseille region of interest toolbox for SPM) will be used for ROI analysis.

Neurofeedback sessions Participants will undergo 10 H.E.G. sessions, twice weekly, over 5 weeks of intervention. They will be instructed to come to sessions in a "half-satiated" condition in order to focus on hedonic/emotional brain circuits involved in eating behavior rather than physiological circuits, based on the "real", physiological hunger. Participants will be given introspective tasks of mindfulness, increased sense of self-control and reduced food craving and will be instructed to attempts augmentation for visual feedback. These tasks correlate with modulation of our ROIs: Increase self-control - is adjusted to increase activity in the superior orbitofrontal cortex (sOFC) whereas suppressing food craving is adjusted to modification of neural activity in the anterior cingulated cortex (ACC) bilaterally. Successive feedback regarding changes in activity in this region will be given analogically with a thermometer with bars above baseline level of activation colored in red while those below baseline colored blue. Thermometer bars are constantly updated with a minimal inherent delay.

ELIGIBILITY:
Inclusion Criteria:

Right handed BMI in the range of 28-35kg/m2

Exclusion Criteria:

* Current or past history of any major psychiatric disorder
* Major medical or neurological disorders
* Exposure to drugs likely to influence cerebral blood flow or neurological function within 3 weeks
* History of drug or alcohol abuse
* General MRI exclusion criteria

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Estimated)
Dates: Start 2015-06; Primary Completion 2015-10 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Increase brain activity in frontal brain areas | 7 weeks

SECONDARY OUTCOMES:
Increased activation of superior frontal brain regions and middle temporal regions in response to food stimuli, in the second fMRI session, perforemed after the neurofeedback sessions, compared to baseline session | 7 weeks
  Activation of superior frontal brain regions and middle temporal regions in response to food stimuli, known to correlate with inhibition, self control and executive functions.
Behavioural measures | 12 months
  Increased scores of self control and inhibition and decreased scores of binge eating and emotional eating on questionnaires.
Anthropometric measures | 12 months
  weight loss according to follow-up 6 and 12 months after intervention.
Number of participants with adverse events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Percik, MD, Principal Investigator — Sheba Medical Center

REFERENCES:
- [Derived] Percik R, Cina J, Even B, Gitler A, Geva D, Seluk L, Livny A. A pilot study of a novel therapeutic approach to obesity: CNS modification by N.I.R. H.E.G. neurofeedback. Clin Nutr. 2019 Feb;38(1):258-263. doi: 10.1016/j.clnu.2018.01.023. Epub 2018 Feb 15. PMID 29428788